CLINICAL TRIAL: NCT05274945
Title: Total Neoadjuvant Therapy Versus Standard Neoadjuvant Chemoradiation for Locally Advanced Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 122019
Record Dates: First submitted 2022-01-07; First posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-01

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Radiotherapy; Consolidation Chemotherapy; Low Density Lipoprotein Receptor-Related Protein-1; Proctectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- total neoadjuvant therapy (Experimental): patients will be treated by total neoadjuvant therapy, including concurrent chemoradiotherapy in the form of radiotherapy 45 Gy/ 25 fractions then boost 5.4 Gy/3 fractions with concurrent bolus 5-fluorouracil + Calcium leucoverin for first 4 days and last 3 days of radiotherapy or capecitabine at 825 mg\m2 twice daily. Then, after 2-3 weeks preoperative chemotherapy will be started in the form of 6 cycles of FOLFOX or CAPOX. Then, after 3-4 weeks surgery will be done.
  Interventions: Radiation: Radiotherapy; Drug: consolidation chemotherapy; Procedure: TME or APR
- standard neoadjuvant therapy (Active Comparator): patients will be treated by standard neoadjuvant therapy , including concurrent chemoradiotherapy in the form of radiotherapy 45 Gy/ 25 fractions then boost 5.4 Gy/3 fractions with concurrent bolus 5-fluorouracil + Calcium leucoverin for first 4 days and last 3 days of radiotherapy or capecitabine at 825 mg\m2 twice daily . Then, after 6-8 weeks surgery will be performed followed by adjuvant chemotherapy.
  Interventions: Radiation: Radiotherapy; Procedure: TME or APR

INTERVENTIONS:
Radiation: Radiotherapy — radiotherapy 45 Gy/ 25 fractions then boost 5.4 Gy/3 fractions with concurrent bolus 5-fluorouracil
  Other Names: Radiation therapy
Drug: consolidation chemotherapy — 6 cycles of FOLFOX or CAPOX
  Other Names: CTX
  Arms: total neoadjuvant therapy
Procedure: TME or APR — total mesorectal excision or abdominoperineal resection
  Other Names: proctectomy

SUMMARY:
The National Comprehensive Cancer Network (NCCN) guidelines recommend trimodality treatment for patients with middle and low LARC with neoadjuvant chemoradiotherapy (NA-CRT), surgical resection with TME, plus additional chemotherapy (CT), in the adjuvant setting. This has markedly reduced pelvic local recurrence from historically about 25% to about 5-10%. However, the 5-year distant relapse is approximately 30% and continues to be the major cause of rectal cancer death.

One strategy to address this issue is to deliver induction chemotherapy before surgery. Induction chemotherapy may be associated with better treatment compliance and may enable full systemic doses of chemotherapy to be delivered.

The above cited considerations, plus favorable data from preliminary reports exploring this strategy, provides a solid rationale for shifting systemic treatment earlier into the treatment paradigm. The current study will evaluate the efficacy and the safety of total neoadjuvant therapy with standard neoadjuvant chemoradiotherapy for locally advanced rectal cancer patients as regards effects on tumor downstaging, pathological complete response, surgical difficulty and early functional outcome.

DETAILED DESCRIPTION:
Colorectal cancer is the third most commonly diagnosed cancer and the third leading cause of cancer death in men and women in the USA.

Surgery using the total mesorectal excision (TME) remains the cornerstone of curative therapy for patients with nonmetastatic, locally advanced middle and low rectal cancer (LARC).

The National Comprehensive Cancer Network (NCCN) guidelines recommend trimodality treatment for patients with middle and low LARC with neoadjuvant chemoradiotherapy (NA-CRT), surgical resection with TME, plus additional chemotherapy (CT), in the adjuvant setting.

This has markedly reduced pelvic local recurrence from historically about 25% to about 5-10%. However, the 5-year distant relapse is approximately 30% and continues to be the major cause of rectal cancer death.

Several other trials have attempted to demonstrate the benefits of postoperative chemotherapy as an adjunct to preoperative radiation and surgery. These trials either failed to demonstrate an advantage, or were closed early due to poor accrual. One common theme among these trials is poor compliance with adjuvant chemotherapy. Completion rates for planned chemotherapy ranged from 43 to 74% in these trials.

The current rectal cancer treatment might lead to delay in the initiation of adjuvant chemotherapy especially in patients with postoperative complications, and this delay is theoretically disadvantageous in that it allows a window for growth of distant micrometastases which may already exist.

One strategy to address this issue is to deliver induction chemotherapy before surgery. Induction chemotherapy may be associated with better treatment compliance and may enable full systemic doses of chemotherapy to be delivered.

Other theoretical advantage of induction chemotherapy includes the possibility of shrinking or downstaging a locally advanced tumor, thereby facilitating more effective local treatment.

Initial chemotherapy also permits delivery of chemotherapy agents directly to the primary tumor while it has a fully intact vasculature, undisrupted by radiation or surgery.

It was supposed that increased chemoradiation-to-surgery interval would result in increased fibrosis and surgical difficulty.However, previous studies showed no increase in the technical difficulty of the operation with total neoadjuvant therapy.

The above cited considerations, plus favorable data from preliminary reports exploring this strategy, provides a solid rationale for shifting systemic treatment earlier into the treatment paradigm. The current study will evaluate the efficacy and the safety of total neoadjuvant therapy with standard neoadjuvant chemoradiotherapy for locally advanced rectal cancer patients as regards effects on tumor downstaging, pathological complete response, surgical difficulty and early functional outcome.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of rectal cancer
* Inferior margin within 12 cm from the anal verge
* staging must be T3-4,N0 or any T, N +ve

Exclusion Criteria:

* Recurrent or metastatic disease.
* Rectal cancer on top of IBD.
* Hereditary non-polyposis colorectal cancer (HNPCC), or hereditary rectal cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
pathological assessment of response to treatment | 10 days
  The histological sections will be reviewed by the same pathologists and the regression grade will be quantified according to Mandard tumor regression grade with sore 1 representing complete response with no viable tumor cells to score 5 representing no regression.

SECONDARY OUTCOMES:
adverse events of chemotherapy | 6 months
  clinical and laboratory follow up to detect hematological and non hematological adverse effects of chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Samir Ashoor, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No